CLINICAL TRIAL: NCT07041138
Title: Effect of a Multidimensional Intervention Programme on Post-stroke Fatigue
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shamay Ng, Prof, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBTPT
Record Dates: First submitted 2025-06-11; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cognitive behavioural programme with physical training (Experimental)
  Interventions: Behavioral: cognitive behavioural programme with physical training
- health education with physical training (Active Comparator)
  Interventions: Behavioral: health education with physical training
- Usual care (Other)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: cognitive behavioural programme with physical training — Participants will receive 7 sessions of cognitive behavioural programme over 8 weeks and have physical training at home for 8 weeks.
  Arms: cognitive behavioural programme with physical training
Behavioral: health education with physical training — Participants will receive 7 sessions of health education over 8 weeks and have physical training at home for 8 weeks.
  Arms: health education with physical training
Behavioral: Usual Care — Participants will maintain their usual life and activities for 8 weeks.
  Arms: Usual care

SUMMARY:
This study aims to evaluate the effects of a multidimensional intervention programme on fatigue and related outcomes among people with stroke.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with stroke at least 6 months ago
* Fatigue Assessment Scale score ≥20
* cognitively intact

Exclusion Criteria:

* Unstable medical conditions
* with any other neurological diseases

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Fatigue Assessment Scale | baseline, end of week 4, end of week 8, and 3-month after the completion of the intervention
  The scale scores range from 10-50, with higher score indicating higher level of fatigue.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | baseline, end of week 4, end of week 8, and 3-month after the completion of the intervention
  The scale scores range from 0-21, with higher score indicating poorer sleep quality.
Geriatric Depression Scale | baseline, end of week 4, end of week 8, and 3-month after the completion of the intervention
  The scale scores range from 0-15, with higher score indicating worse depressive symptoms.
6-minute walk test | baseline, end of week 4, end of week 8, and 3-month after the completion of the intervention
Cardio-ankle vascular index | baseline, end of week 4, end of week 8, and 3-month after the completion of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No